CLINICAL TRIAL: NCT05641597
Title: Functional Impact of Postoperative Vascularized Free Fibula Flap Harvesting Repair Surgery. Prospective Pilot Study
Brief Title: Functional Impact of Reconstructive Surgery by Harvesting a Vascularized Free Fibula Flap Postoperatively.
Acronym: FIBULAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GUILLIER AOI 2021
Record Dates: First submitted 2022-11-23; First posted 2022-12-07 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Bone Reconstruction by Free Fibula Flap
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Actimetric measurement — Evaluation during 7 days "in real life condition Carried out during the pre-operative evaluation (M0), the post-operative evaluation (M1) and the post-operative evaluation (M6)
Other: Evaluation of plantar flexion, dorsal flexion and ankle eversion forces — Performed at the preoperative (M0), postoperative (M1) and postoperative (M6) assessments
Other: Assessment of static and dynamic balance and quality of life — Performed at the preoperative (M0), postoperative (M1) and postoperative (M6) assessments
Other: Functional gait assessment (TM6) — Performed at the preoperative (M0), postoperative (M1) and postoperative (M6) assessments

SUMMARY:
The fibula is a leg bone that can be used in complex bone reconstruction by reconstructive surgery. This innovative surgical procedure is increasingly used in complex facial (mandibular) reconstructions following cancer and trauma involving a bone segment. Following this surgery, chronic pain and post-operative complications can occur, with a functional impact on locomotion, leading to instability, ankle stiffness and a risk of falls. The causes of functional deficits following surgery remain complex and difficult to objectivate by clinical examination alone. However, these deficits need to be better evaluated to develop specific therapeutic targets that will allow the implementation of a personalized postoperative rehabilitation. At present, no study has been performed to objectively quantify the short- and medium-term functional repercussions of the operation.

This study proposes, for the first time, to quantify the repercussions on muscular and locomotor functions as well as the quality of life after reconstructive surgery by transfer of a free vascularized fibula flap in the short and medium term (1 month and 6 months postoperatively).

This is a biomedical, interventional study, which will take place on the Technological Investigation Platform (PIT) located on the garden level of the Rehabilitation Center (C2R) of the Dijon Bourgogne University Hospital, 35 participants will be included in this study over a period of 36 months. For this study, you will be followed for about 7 months, during 3 obligatory visits

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for bone reconstruction with a free fibula flap
* Age ≥ 18 years
* Procedure scheduled in the plastic and maxillofacial surgery department of the Dijon University Hospital
* Willingness to comply with the protocol requirements
* Person having given oral, free and informed consent

Exclusion Criteria:

* Person who is not affiliated or not a beneficiary of a social security system
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant, parturient or breastfeeding woman
* Major who is incapable or unable to give oral consent
* Minor
* Indication for bone reconstruction of a lower limb (e.g. femur) or pelvis
* Musculoskeletal or neurological disorders causing significant prior impairment of walking (whatever the etiology)
* Cognitive disorders that prevent the proper understanding of instructions and the completion of questionnaires
* Non operated patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum isometric force of plantar flexion of the foot on a dynamometer | Change from pre-op and 6 months post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France